CLINICAL TRIAL: NCT03686969
Title: Double-blind, Randomized, Placebo-Controlled Phase III Study Evaluating Efficacy and Safety of Subcutaneous Human Immunoglobulin (Octanorm) in Patients With Dermatomyositis (SCGAM-02)
Brief Title: Study Evaluating Efficacy and Safety of Octanorm in Patients With Dermatomyositis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study complexity, low study recruitment
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCGAM-02
Record Dates: First submitted 2018-08-31; First posted 2018-09-27 (Actual); Results first posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Octanorm (Experimental): 0.5g/kg/week octanorm 16.5%
  Interventions: Drug: Octanorm
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Octanorm — Octanorm 0.5g/kg/week
  Arms: Octanorm
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED PHASE III STUDY EVALUATING EFFICACY AND SAFETY OF SUBCUTANEOUS HUMAN IMMUNOGLOBULIN (OCTANORM) IN PATIENTS WITH DERMATOMYOSITIS

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with diagnosis of definite or probable DM according to the Bohan and Peter criteria.
2. Subjects who have responded to IGIV treatment as assessed by the treating physician and being on a stable dose for at least 3 months on 2 g/kg bodyweight (+/- 10%).
3. For subjects being on other medication(s) for the treatment of DM (immunosuppressants, corticosteroids): a) subject was on such medication(s) at the start of IGIV treatment in the first place, and b) received such medication(s) for at least 3 months prior to study enrolment and at a stable dose for at least 4 weeks prior to study enrolment at the maximally allowed conditions as per Table 2 (see section 4.2.1).
4. MMT-8 score ≥144, with at least 3 other CSM to be normal or near normal as per the following criteria: Visual Analogue Scale [VAS] of patient global disease activity ≤2 cm, physician's global disease activity ≤2 cm, extra-muscular disease activity ≤2 cm; no muscle enzyme >4 times upper limit of normal due to myositis, Health Assessment Questionnaire [HAQ] ≤0.25.
5. Males or females ≥ 18 to <80 years of age.
6. Voluntarily given, fully informed written consent obtained from subject before any study-related procedures are conducted.
7. Subject must be capable and willing to understand and comply with the relevant aspects of the study protocol.

Exclusion Criteria:

1. Cancer-associated myositis, defined as the diagnosis of myositis within 2 years of the diagnosis of cancer (except basal or squamous cell skin cancer or carcinoma in situ of the cervix that has been excised and cured and at least 1 or 5 years, respectively, have passed since excision).
2. Evidence of active malignant disease or malignancies diagnosed within the previous 5 years (including hematological malignancies and solid tumors) or breast cancer diagnosed within the previous 10 years. Subjects >5 years (>10 years for breast cancer) of cancer diagnosis who have been treated and are in remission are allowed.
3. Subjects with overlap myositis (except for overlap with Sjögren's syndrome), connective tissue disease associated DM, inclusion body myositis, polymyositis or drug-induced myopathy.
4. Subjects with immune-mediated necrotizing myopathy with absence of typical DM rash.
5. Subjects with generalized, severe musculoskeletal conditions other than DM that prevent a sufficient assessment of the subject by the physician.
6. Subjects who received blood or plasma-derived products (other than IGIV) or plasma exchange within the last 3 months before enrolment.
7. Subjects with administration of permitted concomitant medications exceeding the maximally allowed conditions as per section 4.2.1.
8. Subjects with administration of forbidden concomitant medications within the washout periods as defined in Table 3: see section 4.2.2.
9. Subjects starting or planning to start a physical therapy-directed exercise regimen during the trial. Subjects on stable physical therapy for >4 weeks are allowed but the regimen should remain the same throughout the trial.
10. Cardiac insufficiency (New York Heart Association III/IV), cardiomyopathy, significant cardiac dysrhythmia requiring treatment, unstable or advanced ischemic heart disease.
11. Severe liver disease, with signs of ascites and hepatic encephalopathy.
12. Severe kidney disease (as defined by estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2).
13. Known hepatitis B, hepatitis C or HIV infection.
14. Subjects with a history of deep vein thrombosis within the last year prior to study enrolment or pulmonary embolism ever.
15. Body mass index >40 kg/m2 and/or body weight >120 kg.
16. Medical conditions whose symptoms and effects could alter protein catabolism and/or IgG utilization (e.g. protein-losing enteropathies, nephrotic syndrome).
17. Known IgA deficiency with antibodies to IgA.
18. History of hypersensitivity, anaphylaxis or severe systemic response to immunoglobulin, blood or plasma derived products or any component of octanorm 16.5% such as polysorbate 80 or to sodium chloride.
19. Known blood hyperviscosity, or other hypercoagulable states.
20. Subjects with a history of drug abuse within the past 5 years prior to study enrolment.
21. Participating in another interventional clinical study with investigational treatment within 3 months prior to study enrolment. Subjects who participated in the Octagam 10% Dermatomyositis Study (GAM10-08) can be included.
22. Women who are breast feeding, pregnant, or planning to become pregnant, or are unwilling to apply an effective birth control method (as per protocol section 7.3.9 b) up to four weeks after the last IMP infusion received.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2018-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- I.M. SECHENOV FIRST MOSCOW STATE MEDICAL UNIVERSITY Rheumatology Department Of, Clinici Of Nephrology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Octanorm | Placebo
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Study terminated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Early study termination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Octanorm | Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Customized [Number; unit: years]
  Age | 52 |  | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: MMT-8
Description: MMT-8; a set of 8 designated muscles tested bilaterally [potential score 0 - 150]
Time Frame: 32 weeks
Population: The study was terminated prematurely. Due to the limited data available (only one patient enrolled and treated), efficacy and safety analyses were not performed.
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: CDASI
Description: The CDASI is a clinician-scored single page instrument that separately measures activity and damage in the skin of DM patients for use in clinical practice or clinical/therapeutic studies.
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Physician's Global Disease Activity VAS Worsening
Description: Physician's Global Disease Activity (10 cm VAS assessing global disease activity from "No evidence of disease activity" to "Extremely active or severe disease activity"; Disease Activity being defined as potentially reversible pathology or physiology resulting from the myositis).
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Extra-Muscular Disease Activity
Description: Extra-muscular activity (part of MDAAT; a combined tool that captures the physician's assessment of disease activity of various organ systems using a scale from 0 = "Not present in the last 4 weeks" to 4 = "New - in the last 4 weeks [compared to the previous 4 weeks]" and a VAS).
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Muscle Enzymes - Aldolase
Description: Measurement of aldolase in blood
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Muscle Enzymes - Creatine Kinase
Description: Measurement of creatine kinase in blood
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Muscle Enzymes - Alanine Aminotransferase
Description: Measurement of alanine aminotransferase in blood
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Muscle Enzymes - Aspartate Aminotransferase
Description: Measurement of aspartate aminotransferase in blood
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Muscle Enzymes - Lactate Dehydrogenase
Description: Measurement of lactate dehydrogenase in blood
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Health Assessment Questionnaire
Description: • Health Assessment Questionnaire (HAQ; a generic rather than a disease-specific instrument; comprised of 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are 2 or 3 questions for each section. Scoring within each section is from 0 [without any difficulty] to 3 [unable to do]. For each section the score given to that section is the worst score within the section. The 8 scores of the 8 sections are summed and divided by 8).
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: SF-36v2 Health Survey
Description: The SF-36 is a multi-purpose, short-form health survey with only 36 questions. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index.
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Mean Change in TIS
Description: Total Improvement Score
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Time to Clinically Important Deterioration
Description: Time to clinically important deterioration
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Adverse Events
Description: Occurrence of all adverse events
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: TEEs
Description: Monitoring safety with occurrence of all thromboembolic events (TEEs)
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: HTRs
Description: Monitoring safety with occurrence of all hemolytic transfusion reactions (HTRs)
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Injection Site Reactions
Description: Monitoring safety by assessing local injection site reactions
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Blood Pressure
Description: Monitoring safety through blood pressure values
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Heart Rate
Description: Monitoring safety through heart rate values
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Body Temperature
Description: Monitoring safety through body temperature values
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Respiratory Rate
Description: Monitoring safety through respiratory rate values
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Physical Examination
Description: The physical examination outcome will be analyzed based on changes from baseline as adverse events.
Time Frame: 32 Weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Sodium
Description: Monitoring safety through lab sodium levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Potassium
Description: Monitoring safety through lab potassium levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Glucose
Description: Monitoring safety through lab glucose levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: ALAT
Description: Monitoring safety through lab ALAT levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: ASAT
Description: Monitoring safety through lab ASAT levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: LDH
Description: Monitoring safety through lab LDH levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Total Bilirubin
Description: Monitoring safety through lab total bilirubin levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Blood Urea Nitrogen
Description: Monitoring safety through lab blood urea nitrogen levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Urea
Description: Monitoring safety through lab urea levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Creatinine
Description: Monitoring safety through lab creatinine levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Albumin
Description: Monitoring safety through lab albumin levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Hematocrit
Description: Monitoring safety through lab hematocrit levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Hemoglobin
Description: Monitoring safety through lab hemoglobin levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

36. Secondary Outcome: Red Blood Cell Count
Description: Monitoring safety through lab red blood cell count levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

37. Secondary Outcome: White Blood Cell Count
Description: Monitoring safety through lab white blood cell count levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

38. Secondary Outcome: Platelets
Description: Monitoring safety through lab platelet levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: Serum Haptoglobin
Description: Monitoring safety through lab serum haptoglobin levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

40. Secondary Outcome: Plasma-Free Hemoglobin
Description: Monitoring safety through lab plasma-free hemoglobin
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

41. Secondary Outcome: Direct Coombs' Test
Description: Monitoring safety through Direct Coombs' test
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

42. Secondary Outcome: D-dimers
Description: Monitoring safety through D-dimers test
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

43. Secondary Outcome: Serum IgG
Description: Monitoring safety through lab IgG levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

44. Secondary Outcome: Aldolase
Description: Monitoring safety through lab aldolase levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

45. Secondary Outcome: Creatine Kinase
Description: Monitoring safety through lab creatine kinase levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

46. Secondary Outcome: Pregnancy Test
Description: Monitoring safety through pregnancy test
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

47. Secondary Outcome: Urine Protein
Description: Monitoring safety through lab urine protein levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

48. Secondary Outcome: Urine Glucose
Description: Monitoring safety through lab urine glucose levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

49. Secondary Outcome: Urine pH
Description: Monitoring safety through lab urine pH levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

50. Secondary Outcome: Urine Nitrite
Description: Monitoring safety through lab urine nitrite levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

51. Secondary Outcome: Urine Ketones
Description: Monitoring safety through lab urine ketone levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

52. Secondary Outcome: Urine Leukocytes
Description: Monitoring safety through lab urine leukocyte levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

53. Secondary Outcome: Urine Hemoglobin
Description: Monitoring safety through lab urine hemoglobin levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

54. Secondary Outcome: Urine Bilirubin
Description: Monitoring safety through lab urine bilirubin levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

55. Secondary Outcome: Urine Urobilinogen
Description: Monitoring safety through lab urine urobilinogen levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

56. Secondary Outcome: Urine Hemosiderin
Description: Monitoring safety through lab urine hemosiderin levels
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

57. Secondary Outcome: HIV
Description: Monitoring safety through HIV testing
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

58. Secondary Outcome: Hepatitis B
Description: Monitoring safety through hepatitis B testing
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

59. Secondary Outcome: Hepatitis C
Description: Monitoring safety through hepatitis C testing
Time Frame: 32 weeks
Population: as for outcome 1
Arm/Group | Octanorm | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The patient was treated according to the protocol until week 14 Treatment after week 14 was discontinued because of early study termination
Description: Number of patients at risk for SAEs, All-Cause Mortality, and other adverse events in placebo group is 0 as 0 patients were enrolled into the placebo group.
Arm/Group | Octanorm | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octanorm (N=1) | Placebo (N=0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (2) | NA
Infusion site haematoma (General disorders) | 1 (1) | NA
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | NA
Blood creatine phosphokinase increased (Investigations) | 1 (1) | NA
Aldolase increased (Investigations) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT03686969/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT03686969/SAP_001.pdf